CLINICAL TRIAL: NCT05039398
Title: A Policy Developed Intervention With Additional Participatory Dialogue and Guidance for Improved Occupational Health and Safety (OHS) Among Workplaces With WEA (Working Environment Authority) Violations
Brief Title: 'Dialogue and Guidance' - a Policy Intervention for Improved OHS Among Workplaces With WEA Violations
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Danish Labor Inspectorate (Other Government)
Collaborators: National Research Centre for the Working Environment, Denmark (Other Government)
Responsible Party: Principal Investigator, Johan Simonsen Abildgaard, Senior Researcher, National Research Centre for the Working Environment, Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AT-D&V
Record Dates: First submitted 2021-06-01; First posted 2021-09-09 (Actual); Last update posted 2021-09-09 (Actual); Status verified 2021-09

CONDITIONS: Occupational Diseases; Occupational Injuries; Safety Issues
MeSH Terms: conditions — Occupational Diseases; Occupational Injuries | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Parallel Assignment Each workplace assigned for inspection by the WEA is randomized to either of two intervention groups (physical meeting dialogue and guidance, telephone meeting dialogue and guidance) or a control group. If the workplace receives a WEA notice of material violations of work environment regulations, the workplace receives an offer for dialogue and guidance if they are in one of the two intervention groups. The comparison group receives treatment as usual.
  Randomization as follows:
  1/3 are randomized to treatment-as-usual comparison status 1/3 are randomized to receive dialogue and guidance over telephone 1/3 are randomized to receive dialogue and guidance at a physical meeting
Masking Description: None (Open Label) During inspection by the WEA the intervention status is masked for both the inspector and the assessed workplace. After the inspection is complete and all violation notices are sent to the company, the intervention group additionally receives invitation to a dialogue and guidance meeting. From this point the intervention is not masked.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Comparison group (Active Comparator)
  Interventions: Behavioral: Treatment as usual
- Telephone D&G (Experimental)
  Interventions: Behavioral: Dialogue and guidance over telephone
- Physical meeting D&G (Experimental)
  Interventions: Behavioral: Dialogue and guidance at physical meeting

INTERVENTIONS:
Behavioral: Treatment as usual — The workplace receives dialogue and guidance during the WEA workplace inspection as per WEA standard practice.
  Arms: Comparison group
Behavioral: Dialogue and guidance over telephone — In addition to receiving dialogue and guidance during WEA workplace inspection as standard practice by the WEA, the "Dialogue and guidance over telephone" receives up to 2 hours of supplemental dialogue and guidance after WEA inspection with the WEA inspector. This is conducted over the telephone.
  Arms: Telephone D&G
Behavioral: Dialogue and guidance at physical meeting — In addition to receiving dialogue and guidance during WEA workplace inspection as standard practice by the WEA, the "Dialogue and guidance at physical meeting" receives up to 2 hours of supplemental dialogue and guidance after WEA inspection with the WEA inspector. This is conducted as a physical meeting.
  Arms: Physical meeting D&G

SUMMARY:
With the aim to inspire and motivate workplaces in their work to prevent and reduce occupational health and safety hazards, the Danish Working Environment Authority (WEA) developed the intervention 'Dialogue and Guidance' aimed at workplaces receiving notices (prohibition notice, immediate improvement notice and notice with time limit) from WEA during inspections. At present, WEA gives dialogue and guidance as standard practice during WEA inspections to all workplaces receiving a notice with the purpose to help workplaces resolve the occupational health and safety problem that led to the notice. In the intervention 'Dialogue and Guidance' the experimental groups are receiving additional dialogue and guidance at a subsequent meeting (over the telephone or physical presence) that takes place after the inspection and after the deadline for appealing the notice has expired. The control group is receiving dialogue and guidance during inspection as usual.

The aim of this RCT study is to evaluate the policy-developed intervention with additional 'Dialogue and Guidance' in regards to the effect on motivation and priority of occupational health and safety work at the workplace after 6 months follow-up and for WEA notices by next WEA inspection (approx. follow-up by 12-18 months).

Study is risk assessed and approved under Danish Data Protection Agency via the National Research Centre for the Working Environment's umbrella approval.

ELIGIBILITY:
Subjects under inspection are workplaces, and respondents of the questionnaires are the workplace manager and a work environment representative or shop steward.

Inclusion Criteria:

• Workplaces (production units) who receives a WEA notice during WEA inspection through the period of intervention. The following WEA notices are included:

* Immediate improvement notice
* Notice with time limit (material)

Exclusion Criteria:

* Companies with 0-1 employees.
* Production units from the construction industry met on temporary worksites (such as construction sites) that have more than one employee and does not have a certified occupational health and safety management system.
* Companies receiving notices only about issues in the formal/procedural aspects of the work environment (such as flaws in the workplace risk assessment) and no other notices.
* Companies receiving more than four reactions from WEA at the inspection (as these receive a competency notice and are not included in the study).
* Companies that receive a prohibition notice by the WEA inspector due to severity of work environment violations.
* A WEA improvement notice is not eligible for inclusion in the study if the workplace has entered into a collaborative agreement with WEA on improvement of the issue, or if they have received a competency notice on the WEA issue.
* Companies receiving WEA inspections in relation to initiatives targeting social dumping

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4500 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
WEA notices - specific | Through study completion, approx. 12-18 months
  Change from baseline WEA inspection in number of WEA notices of the same specific type (topic-code specific) at next WEA inspection (approx. 12-18 months after).
  WEA notices included for study:
  1. prohibition notice (+ topic-code)
  2. immediate notice (+ topic-code)
  3. notice with time limit (+ topic-code)
  Register data provided by the Danish Labour Authority
  (Intervention is hypothesized to lead to fewer notices)
WEA notices - all | Through study completion, approx. 12-18 months
  Change from baseline WEA inspection in number of received WEA notices at next WEA inspection (approx. 12-18 months after).
  WEA notices included for study:
  1. prohibition notice (all)
  2. immediate notice (all)
  3. notice with time limit (all)
  Register data provided by the Danish Labour Authority
  (Intervention is hypothesized to lead to fewer notices)
OHS problem solution | Baseline to 6 months follow-up
  Comparison of item score between intervention groups and comparison group on the following:
  • One single item on if they solved the OHS problem that led to WEA notice (response categories: yes, no, partially).
  (Intervention is hypothesized to lead to higher rates of having solved the OHS problems in question)
Sustainable OHS solutions | Baseline to 6 months follow-up
  Comparison of an index score consisting of two items scored on a 5-point Likert-scale between intervention groups and comparison group on whether the implemented solution to WEA violation has led to sustainable changes in the workplace .
  Sample item: "The implemented OHS solution to solve the WEA violation makes it unlikely that a similar OHS problem will arise in the future" An index score is calculated from the mean of the two items (i.e. the index has a range from 1 to 5) Higher scores equals higher sustainability of OHS solutions.
  (intervention is hypothesized to lead to higher values)

SECONDARY OUTCOMES:
OHS motivation | Baseline to 6 months follow-up
  Comparison of item score between intervention groups and comparison group on three single items related to workplace OHS motivation measured on a 5-point Likert-scale.
  The items are:
  "The employees are very motivated to improve the work environment" "The management is very motivated to improve the work environment" "Working with the OHS solution has made the people involved more motivated to work on OHS problems" Higher scores equals higher OHS motivation.
  (intervention is hypothesized to lead to higher values)
OHS priority | Baseline to 6 months follow-up
  Comparison of scale score between intervention groups and comparison group on the following:
  • Scale measuring OHS priority consisting of three 5-point Likert-scale items from the national workplace-survey 'Work Environment Activities in Danish Workplaces'.
  Sample item: "The workplace prioritizes prevention of OHS problems highly". A scale score is calculated from the mean of the items (i.e. the scale has a range from 1 to 5 ). Higher scores equals higher OHS priority.
  (intervention is hypothesized to lead to higher values)
OHS practice efficacy | Baseline to 6 months follow-up
  Comparison of item score between intervention groups and comparison group on the following:
  • A scale consisting of six 5-point Likert-scale items developed for the D&V-project measuring OHS practice behaviours.
  Sample items include e.g.:
  "We follow up on whether OHS initiatives have the desired effect" "We continuously solve the OHS problems that arise" A scale score is calculated from the mean of the items (i.e. the scale has a range from 1 to 5) Higher scores equals higher OHS practice efficacy.
  (intervention is hypothesized to lead to higher values)
Diffusion of OHS knowledge | Baseline to 6 months follow-up
  Comparison of an index consisting of two items scored on a 5-point Likert-scale between intervention groups and comparison group on whether the knowledge from implemented solution to WEA violation has been spread to other areas/problems.
  Sample item: "We are good at disseminating OHS knowledge in our organization".
  An index score is calculated from the mean of the two items (i.e. the index has a range from 1 to 5) Higher scores equals higher diffusion of OHS solutions.
  (intervention is hypothesized to lead to higher values)
Other WEA reactions | Through study completion, approx. 12-18 months
  Change from baseline WEA inspection in number of other WEA reactions by next WEA inspection (approx. 12-18 months after).
  Other WEA reaction includes the following:
  * Ruling without obligation to act
  * Investigation notice (§ 21 notice)
  * Competence notice
  * Guidance
  (Intervention is hypothesized to lead to fewer reactions)

CONTACTS AND LOCATIONS:
Overall Officials: Johan S. Abildgaard, PhD, Principal Investigator — The National Research Centre for the Working Environment
Locations (1):
- Working Environment Authority, Copenhagen, Copenhagen Ø, Denmark